CLINICAL TRIAL: NCT02670161
Title: Quality Improvement and Practice Based Research in Neurology Using the Electronic Medical Record
Brief Title: Quality Improvement and Practice Based Research in Neurology Using the EMR
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Steven Meyers, Senior Clinician Educator, Department of Neurology, Endeavor Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH14-355; 1R01HS024057-01 (AHRQ)
Record Dates: First submitted 2016-01-23; First posted 2016-02-01 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Brain Tumors; Epilepsy; Migraine; Mild Cognitive Impairment; Concussion; Multiple Sclerosis; Neuropathy; Parkinson's; Restless Legs Syndrome; Stroke
MeSH Terms: conditions — Brain Neoplasms; Epilepsy; Migraine Disorders; Cognitive Dysfunction; Brain Concussion; Multiple Sclerosis; Parkinson Disease; Restless Legs Syndrome; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (see interventions description) (Active Comparator): The investigators will conduct 11 pragmatic trials using the EMR: brain tumors (prevent seizures), epilepsy (prevent other seizure types), mild cognitive impairment (improve memory), migraine (prevention), migraine (abortive), mild traumatic brain injury (prevent post concussion syndrome), multiple sclerosis (attenuate relapses), neuropathy (pain management), Parkinson's (treat motor symptoms), restless legs syndrome (treat sensory symptoms), stroke (secondary prevention). For each trial they will compare up to three medications or treatments either FDA approved for the indication, or commonly employed. The pragmatic trials will be small and primarily to demonstrate the feasibility of subgroup based adaptive assignment of treatments, electronic consenting, and data capture at the point of care using the EMR. The focus is on the development of the study design and methodology and not on the treatments per se.
  Interventions: Drug: Listed for each disorder below, up to three drugs per disorder (too many characters to list in this field; see Intervention Description)
- Treatment B (see interventions description) (Active Comparator): The investigators will conduct 11 pragmatic trials using the EMR: brain tumors (prevent seizures), epilepsy (prevent other seizure types), mild cognitive impairment (improve memory), migraine (prevention), migraine (abortive), mild traumatic brain injury (prevent post concussion syndrome), multiple sclerosis (attenuate relapses), neuropathy (pain management), Parkinson's (treat motor symptoms), restless legs syndrome (treat sensory symptoms), stroke (secondary prevention). For each trial they will compare up to three medications or treatments either FDA approved for the indication, or commonly employed. The pragmatic trials will be small and primarily to demonstrate the feasibility of subgroup based adaptive assignment of treatments, electronic consenting, and data capture at the point of care using the EMR. The focus is on the development of the study design and methodology and not on the treatments per se.
  Interventions: Drug: Listed for each disorder below, up to three drugs per disorder (too many characters to list in this field; see Intervention Description)
- Treatment C (see interventions description) (Active Comparator): The investigators will conduct 11 pragmatic trials using the EMR: brain tumors (prevent seizures), epilepsy (prevent other seizure types), mild cognitive impairment (improve memory), migraine (prevention), migraine (abortive), mild traumatic brain injury (prevent post concussion syndrome), multiple sclerosis (attenuate relapses), neuropathy (pain management), Parkinson's (treat motor symptoms), restless legs syndrome (treat sensory symptoms), stroke (secondary prevention). For each trial they will compare up to three medications or treatments either FDA approved for the indication, or commonly employed. The pragmatic trials will be small and primarily to demonstrate the feasibility of subgroup based adaptive assignment of treatments, electronic consenting, and data capture at the point of care using the EMR. The focus is on the development of the study design and methodology and not on the treatments per se.
  Interventions: Drug: Listed for each disorder below, up to three drugs per disorder (too many characters to list in this field; see Intervention Description)

INTERVENTIONS:
Drug: Listed for each disorder below, up to three drugs per disorder (too many characters to list in this field; see Intervention Description) — brain tumors (lamotrigine, levetiracetam, valproic acid), epilepsy (lamotrigine, levetiracetam, valproic acid), mild cognitive impairment (donepezil, rivastigmine, memantine), migraine (amitriptyline, propranolol, topiramate), migraine (sumatriptan, rizatriptan, zolmitriptan), mild traumatic brain injury (omega-3 fatty acids, education only), multiple sclerosis (ACTH, methylprednisolone), neuropathy (duloxetine, pregabalin, amitryptiline), Parkinson's disease (pramipexole, ropinerole, rotigotine), restless legs syndrome (pramipexole, ropinerole, rotigotine), stroke (aspirin, clopidogrel).
  Other Names: (too many characters to list in this field; see Intervention Description)

SUMMARY:
The investigators will conduct at NorthShore University HealthSystem pragmatic trials using the EMR for 10 common neurological disorders. They will demonstrate the feasibility of subgroup based adaptive assignment of treatments, electronic consenting, and outcomes data capture at the point of care using the EMR. They will identify the most effective treatments for common neurological disorders and seek replication by the NPBRN.

DETAILED DESCRIPTION:
The goals of the proposed research are to advance quality improvement and practice based research in Neurology using the electronic medical record (EMR). The American Academy of Neurology (AAN) has published evidence-based guidelines, quality improvement measures, and resources for several neurological disorders. However, the AAN guidelines and measures have not been implemented routinely and benchmark data are lacking. There are few EMR tools available to standardize neurology office visits according to Best Practices, to provide alerts when neurological care is deviating from AAN guidelines, to capture data regarding adherence to AAN or other quality parameters, to measure the effects of compliance with guidelines on outcomes, or to share longitudinal data and to compare effectiveness of care across neurological practices. The Department of Neurology at NorthShore University HealthSystem (NorthShore) has built into its commercial EMR "Epic" structured clinical documentation support (SCDS) and clinical decision support (CDS) tools that standardize care, write progress notes, and capture up to 1,000 discrete and cascading fields of neurological data per office visit. However, these EMR tools have not been disseminated for use by other Neurology practices or for data sharing, and presently do not support clinical trials. Pragmatic trials using EMRs would enable comparisons of treatments at the point of care. To address gaps in quality improvement and practice based research in Neurology, the investigators are proposing to the Agency for Healthcare Research and Quality (AHRQ) a project with the specific aims: 1) To create a Neurology Practice Based Research Network (NPBRN). The NorthShore site will share SCDS and CDS tools for 10 common neurological disorders (brain tumors, epilepsy, migraine, mild cognitive impairment, mild traumatic brain injury, multiple sclerosis, neuropathy, Parkinson's disease, restless legs syndrome, and stroke) with seven other Department of Neurology that also use the Epic EMR platform (eight sites total). 2) To conduct at NorthShore pragmatic trials using the EMR for 10 common neurological disorders. The investigators will demonstrate the feasibility of subgroup based adaptive assignment of treatments, electronic consenting, and outcomes data capture at the point of care using the EMR. They will identify the most effective treatments for common neurological disorders and seek replication by the NPBRN. The aims are innovative because the investigators will use the EMR to hardwire quality and outcomes research in Neurology. They will individualize medicine at the point of care by conducting pragmatic trials using subgroup based adaptive designs, comparing the effectiveness of available treatments for common neurological disorders. The aims are significant because they are studying several neurological disorders, a leading cause of healthcare burden worldwide. They will create a national practice based network to improve health care quality by accelerating implementation of patient-centered outcomes research in Neurology using the EMR, and evidence to make health care safer and to improve health care efficiency. NOTE: This ClinicalTrials.gov registration relates to Aim 2 of the project (pragmatic trials using the EMR). Aim 1 is an observational study only (quality improvement, comparative effectiveness research).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brain tumors, epilepsy, migraine, mild cognitive impairment (concussion), mild traumatic brain injury, multiple sclerosis, neuropathy, Parkinson's disease, restless legs syndrome, and stroke.
* Eligible to receive any of the three compared treatments according to FDA approval for the indication or off label use according to standard of care.

Exclusion Criteria:

-- None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
survival free of discontinuation or alternative prevention drug (migraine trial) | six months
survival free of disability measured by FAQ score 9+ (memory trial) | one year
survival free of discontinuation or alternative anti epileptic drug (epilepsy trial) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maraganore DM, Frigerio R, Kazmi N, Meyers SL, Sefa M, Walters SA, Silverstein JC. Quality improvement and practice-based research in neurology using the electronic medical record. Neurol Clin Pract. 2015 Oct;5(5):419-429. doi: 10.1212/CPJ.0000000000000176. PMID 26576324
- [Background] Narayanan J, Dobrin S, Choi J, Rubin S, Pham A, Patel V, Frigerio R, Maurer D, Gupta P, Link L, Walters S, Wang C, Ji Y, Maraganore DM. Structured clinical documentation in the electronic medical record to improve quality and to support practice-based research in epilepsy. Epilepsia. 2017 Jan;58(1):68-76. doi: 10.1111/epi.13607. Epub 2016 Nov 19. PMID 27864833
- See also: Publication — http://onlinelibrary.wiley.com/doi/10.1111/epi.13607/full
- See also: Project Summary (AHRQ) — https://reporter.nih.gov/project-details/8938766